CLINICAL TRIAL: NCT03646019
Title: Serum Oxidative Status as a Potential Predictor of Coronary Artery Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prof. Tony hayek MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Tony hayek MD, Director, Department of Internal Medicine E, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Other Study IDs: 0373-18-RMB
Record Dates: First submitted 2018-08-10; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Paraoxanase 1; Thiobarbituric Acid Reactive Substances; Thiol Groups
Keywords: Coronary artery disease; paraoxanase 1; Thiobarbituric Acid Reactive Substances; Thiol groups
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal coronary arteries
- Non significant coronary artery disease
- Significant coronary artery disease

SUMMARY:
Coronary artery disease (CAD) is a major cause of death and disability in developed countries.Human studies revealed a significant association between serum oxidative status using PON1, TBARS and thiol levels and the presence of CAD and its severity. However, these studies were addressing the severity of CAD depending on coronary angiography of patients presenting with ST elevation myocardial infarction, Non ST elevation myocardial infarction, unstable angina pectoris, while part of them even had a history of CAD. Others where admitted for an elective coronary angiography for suspected stable CAD while only few patients were assessed for atypical chest pain. This study thus aims to assess the relationship between PON1 activity, TBARS and thiol levels and the existence of CAD and its severity in patients with no previous history of CAD presenting to the emergency department (ED) with acute chest pain but with no evidence of acute myocardial infarction or acute E.C.G ischemic changes. Assessment with a Cardiac CT scan instead of coronary angiography will allow the investigators to study the status of coronary atherosclerosis and calcium burden in all participants, including those presenting with atypical chest pain that most probably will not be referred by physicians to a coronary angiography. Further sub groups analysis will estimate this relationship particularly in low-intermediate risk groups depending on 3 different validated scoring systems - TIMI, GRACE and HEART score.

DETAILED DESCRIPTION:
Oxidized low-density lipoprotein (LDL) has a pivotal role in the initiation as well as the progression of atherosclerosis. High-density lipoprotein (HDL) exerts a protective effect on the cardiovascular system, and serum HDL-cholesterol levels correlates inversely with atherosclerosis severity, since it protects against oxidative damage. It is believed that the anti oxidant activity of HDL is mainly determined by the HDL-associated enzyme paraoxanase 1 (PON1). The direct role of PON1 in reducing oxidative stress was demonstrated in studies using the PON1 knock out mice model and the human PON1 transgenic mice model. HDL particles isolated from PON1-deficient mice were unable to inhibit LDL oxidation in cultured arterial cells, in contrast to the HDL isolated from control mice. Moreover, HDL isolated from PON1 transgenic mice (that exhibited 3-fold increase in PON1 activity) was more effective in protecting LDL against oxidation compared to control / wild type mice. PON1 was shown to inhibit cholesterol influx by reducing the formation of oxidized LDL, increasing the breakdown of specific oxidized lipids in oxidized LDL, and decreasing macrophage uptake of oxidized LDL. PON1 also inhibits cholesterol biosynthesis and stimulates HDL-mediated cholesterol efflux from macrophages. Human studies revealed a significant association between decreased PON1 activity and increased risk of CAD. Mean PON1 activity levels were lower in patients with acute myocardial infarction (AMI) than stable CAD patients and highest level were observed in control patients. In patients with AMI, PON1 activity increased significantly within 6 weeks of the acute event, even though it was still markedly lower as compared to the stable CAD patients. Suggesting that sudden lowering of serum PON1 activity in a population which already has lower activity may be one of the risk factors for development of AMI. Ayub et al. has reported that serum PON1 activity was already decreased within 2 hours of the onset of symptoms of AMI and remained low subsequently, suggesting that the decreased PON1 activity may have preceded the acute event. A prospective study reported that low serum PON1 activity is a predictive risk factor for subsequent coronary events. Moreover, PON1 activity has presented a possible biochemical marker for CAD severity assessed by coronary angiography. Thiobarbituric acid reactive substances (TBARS) is an increased lipid peroxidation indicator that was found to be increased in CAD. A weak but significant correlation was also observed between levels of TBARS and angiographic progression of disease, especially moderate coronary artery stenosis. Elif Azarsiz et al. propose that the elevation in TBARS levels might be a more marked indicator for the degree of atherosclerosis than the insufficiency in antioxidant enzymes such as PON1. Thiol / -SH levels were found to be lower in the CAD group compared with the non CAD group and control group. Decreased serum thiol levels were associated with the presence and severity of CAD.

In this study first set of blood samples will be obtained at presentation to the ED and later on at the department of internal medicine E'in the Rambam's Medical Health Center, including CBC count, creatinine, electrolytes and two high sensitive troponin measurements. A second set of blood samples will be obtained at the morning of the cardiac CT scan after 10-12-h over-night fast, including serum level of HbA1C, CRP, kidney and liver function, total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides. All parameters will be measured on fresh blood samples at the Rambam's Medical Health Center biochemical and endocrine laboratories. Serum oxidative status will be determined by collecting additional blood tube (5 ml of blood) at the morning of the cardiac CT scan. After centrifuging the clotted sample, serum will be separated and stored at minus 40 celsius for further analysis of PON-1 / aryl esterase activity, measurement of protein thiol groups / glutathione and measurement of serum level of thiobarbituric acid reactive substances (TBARS, measured as malondialdehyde [MDA] equivalents), at Lipid Research Laboratory of the Rappaport Faculty of Medicine at the Technion, Haifa - Israel.

Patients not already on beta-blocking drugs will receive oral metoprolol (50-200 mg) for heart rates over 65 beats/min. An additional intravenous metoprolol (5-10 mg) will be administered to achieve a target heart rate <65 beats/min 5-15 minutes before the test. However, no patient will be excluded because of a heart rate above this target.

The cardiac CT scan images will be interpreted by a panel of experienced radiologists blinded to the study, at Rambam Medical Health Center. The degree of coronary obstruction will be measured in terms of the percent of stenosis. Participant with stenosis less than or equal to 49% is considered to have a non significant CAD. Participant with stenosis more than 49% is considered to have a significant CAD. Calcium burden will be measured by the Agatston score. Subjects with significant stenosis in the cardiac CT scan will undergo coronary angiography for a further assessment of the degree of stenosis. Result of the coronary angiography will be assessed in relation to the measurement of serum oxidative status as well.

In this study hypertension will be defined as a DBP ≥ 90 mmHg, SBP ≥ 140 mmHg measured using a calibrated electronic blood pressure machine in both arms while sitting after at least 30 min of rest, and the average of 3 recording will be used or self reported use of anti hypertensive drug. Diabetes mellitus (DM) will be diagnosed if the HbA1C is ≥ 6.5 % or if the patient is treated with insulin or oral hypoglycemic agents. Body mass index (BMI) will be computed as weight /height squared (k/m2).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the chest pain unit (CPU) in the Department of Internal Medicine E' in the Rambam Medical Health center - Israel after they presented to the ED with acute chest pain, suspected to be of cardiac origin and seems to be suitable for further investigation by a cardiac CT scan. Participants will have no previous history of CAD. E.C.G at admission is with no signs of myocardial ischemia and cardiac biomarkers are normal.

Exclusion Criteria:

* known CAD.
* allergy to iodine contrast agents.
* asthma exacerbation.
* current use of steroids or other immunomodulating drugs.
* renal insufficiency (creatinine level ≥ 1.5 mg/dl).
* contraindication for radiations, as in pregnant women.
* fever during the last 48 hours prior to admission.
* concomitant inflammatory diseases (infections, auto immune disorders, kidney and liver diseases, and recent major surgical procedure).
* Subjects with valvular, myocardial or pericardial diseases.
* Poor CT image quality due to motion artifacts or inappropriate contrast delivery, resulting in non-diagnostic image quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the chest pain unit (CPU) in the Department of Internal Medicine E' in the Rambam Medical Health center - Israel after they presented to the ED with acute chest pain, suspected to be of cardiac origin and seems to be suitable for further investigation by a cardiac CT scan. Participants will have no previous history of CAD. E.C.G at admission is with no signs of myocardial ischemia and cardiac biomarkers are normal.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The presence and severity of coronary artery disease assessed by a cardiac CT scan / coronary angiography. | 7 days
  The presence of coronary artery disease is defined as the presence of any atherosclerotic plaque leading to any percentage of coronary artery stenosis. The severity of coronary artery disease is defined either as significant or non significant. A Non significant coronary artery disease is defined as any coronary artery stenosis less than or equal to 49%. A Significant coronary artery disease is defined as any coronary artery stenosis more than 49%.

REFERENCES:
- [Background] Sanchis-Gomar F, Perez-Quilis C, Leischik R, Lucia A. Epidemiology of coronary heart disease and acute coronary syndrome. Ann Transl Med. 2016 Jul;4(13):256. doi: 10.21037/atm.2016.06.33. PMID 27500157
- [Background] Zhou C, Cao J, Shang L, Tong C, Hu H, Wang H, Fan D, Yu H. Reduced paraoxonase 1 activity as a marker for severe coronary artery disease. Dis Markers. 2013;35(2):97-103. doi: 10.1155/2013/816189. Epub 2013 Jul 28. PMID 24167353
- [Background] Rye KA, Barter PJ. Cardioprotective functions of HDLs. J Lipid Res. 2014 Feb;55(2):168-79. doi: 10.1194/jlr.R039297. Epub 2013 Jun 27. PMID 23812558
- [Background] Gur M, Cayli M, Ucar H, Elbasan Z, Sahin DY, Gozukara MY, Selek S, Koyunsever NY, Seker T, Turkoglu C, Kaypakli O, Aksoy N. Paraoxonase (PON1) activity in patients with subclinical thoracic aortic atherosclerosis. Int J Cardiovasc Imaging. 2014 Jun;30(5):889-95. doi: 10.1007/s10554-014-0407-y. Epub 2014 Apr 4. PMID 24700021
- [Background] Singh K, Singh R, Chandra S, Tyagi S. Paraoxonase-1 is a better indicator than HDL of Atherosclerosis - A pilot study in North Indian population. Diabetes Metab Syndr. 2018 May;12(3):275-278. doi: 10.1016/j.dsx.2017.12.006. Epub 2017 Dec 14. PMID 29254890
- [Background] Shih DM, Gu L, Xia YR, Navab M, Li WF, Hama S, Castellani LW, Furlong CE, Costa LG, Fogelman AM, Lusis AJ. Mice lacking serum paraoxonase are susceptible to organophosphate toxicity and atherosclerosis. Nature. 1998 Jul 16;394(6690):284-7. doi: 10.1038/28406. PMID 9685159
- [Background] Shih DM, Xia YR, Wang XP, Miller E, Castellani LW, Subbanagounder G, Cheroutre H, Faull KF, Berliner JA, Witztum JL, Lusis AJ. Combined serum paraoxonase knockout/apolipoprotein E knockout mice exhibit increased lipoprotein oxidation and atherosclerosis. J Biol Chem. 2000 Jun 9;275(23):17527-35. doi: 10.1074/jbc.M910376199. PMID 10748217
- [Background] Oda MN, Bielicki JK, Ho TT, Berger T, Rubin EM, Forte TM. Paraoxonase 1 overexpression in mice and its effect on high-density lipoproteins. Biochem Biophys Res Commun. 2002 Jan 25;290(3):921-7. doi: 10.1006/bbrc.2001.6295. PMID 11798161
- [Background] Tward A, Xia YR, Wang XP, Shi YS, Park C, Castellani LW, Lusis AJ, Shih DM. Decreased atherosclerotic lesion formation in human serum paraoxonase transgenic mice. Circulation. 2002 Jul 23;106(4):484-90. doi: 10.1161/01.cir.0000023623.87083.4f. PMID 12135950
- [Background] Aviram M, Rosenblat M. Paraoxonases 1, 2, and 3, oxidative stress, and macrophage foam cell formation during atherosclerosis development. Free Radic Biol Med. 2004 Nov 1;37(9):1304-16. doi: 10.1016/j.freeradbiomed.2004.06.030. PMID 15454271
- [Background] Zhao Y, Ma Y, Fang Y, Liu L, Wu S, Fu D, Wang X. Association between PON1 activity and coronary heart disease risk: a meta-analysis based on 43 studies. Mol Genet Metab. 2012 Jan;105(1):141-8. doi: 10.1016/j.ymgme.2011.09.018. Epub 2011 Sep 22. PMID 22030099
- [Background] Gocmen AY, Gumuslu S, Semiz E. Association between paraoxonase-1 activity and lipid peroxidation indicator levels in people living in the Antalya region with angiographically documented coronary artery disease. Clin Cardiol. 2004 Jul;27(7):426-30. doi: 10.1002/clc.4960270714. PMID 15298047
- [Background] Ding J, Chen Q, Zhuang X, Feng Z, Xu L, Chen F. Low paraoxonase 1 arylesterase activity and high von Willebrand factor levels are associated with severe coronary atherosclerosis in patients with non-diabetic stable coronary artery disease. Med Sci Monit. 2014 Nov 25;20:2421-9. doi: 10.12659/MSM.890911. PMID 25420483
- [Background] Graner M, James RW, Kahri J, Nieminen MS, Syvanne M, Taskinen MR. Association of paraoxonase-1 activity and concentration with angiographic severity and extent of coronary artery disease. J Am Coll Cardiol. 2006 Jun 20;47(12):2429-35. doi: 10.1016/j.jacc.2006.01.074. Epub 2006 May 26. PMID 16781370
- [Background] Jayakumari N, Thejaseebai G. High prevalence of low serum paraoxonase-1 in subjects with coronary artery disease. J Clin Biochem Nutr. 2009 Nov;45(3):278-84. doi: 10.3164/jcbn.08-255. Epub 2009 Oct 28. PMID 19902017
- [Background] Shekhanawar M, Shekhanawar SM, Krisnaswamy D, Indumati V, Satishkumar D, Vijay V, Rajeshwari T, Amareshwar M. The role of 'paraoxonase-1 activity' as an antioxidant in coronary artery diseases. J Clin Diagn Res. 2013 Jul;7(7):1284-7. doi: 10.7860/JCDR/2013/5144.3118. Epub 2013 Jul 1. PMID 23998046
- [Background] Kuchta A, Strzelecki A, Cwiklinska A, Toton M, Gruchala M, Zdrojewski Z, Kortas-Stempak B, Gliwinska A, Dabkowski K, Jankowski M. PON-1 Activity and Plasma 8-Isoprostane Concentration in Patients with Angiographically Proven Coronary Artery Disease. Oxid Med Cell Longev. 2015;2015:5136937. doi: 10.1155/2016/5136937. Epub 2015 Nov 30. PMID 26697134
- [Background] Cheraghi M, Shahsavari G, Maleki A, Ahmadvand H. Paraoxonase 1 Activity, Lipid Profile, and Atherogenic Indexes Status in Coronary Heart Disease. Rep Biochem Mol Biol. 2017 Oct;6(1):1-7. PMID 29090223
- [Background] Lu C, Gao Y, Zhou H, Tian H. The relationships between PON1 activity as well as oxLDL levels and coronary artery lesions in CHD patients with diabetes mellitus or impaired fasting glucose. Coron Artery Dis. 2008 Dec;19(8):565-73. doi: 10.1097/MCA.0b013e3283109206. PMID 19005291
- [Background] Kaya Z, Salih Aydin M, Hazar A, Can Ata E, Sezen H, Yildiz A, Demirbag R, Aksoy N. Association of serum paraoxonase activity and coronary artery calcification. Eur Rev Med Pharmacol Sci. 2013;17(15):2121-6. PMID 23884836
- [Background] Maturu VN, Gupta N, Singh G, Gill K, Sharma YP, Singh S. Serum Paraoxonase (PON1) Activity in North-West Indian Punjabi's with Acute Myocardial Infarction. Indian J Clin Biochem. 2013 Jul;28(3):248-54. doi: 10.1007/s12291-012-0260-5. Epub 2012 Oct 11. PMID 24426219
- [Background] Ayub A, Mackness MI, Arrol S, Mackness B, Patel J, Durrington PN. Serum paraoxonase after myocardial infarction. Arterioscler Thromb Vasc Biol. 1999 Feb;19(2):330-5. doi: 10.1161/01.atv.19.2.330. PMID 9974415
- [Background] Mackness B, Durrington P, McElduff P, Yarnell J, Azam N, Watt M, Mackness M. Low paraoxonase activity predicts coronary events in the Caerphilly Prospective Study. Circulation. 2003 Jun 10;107(22):2775-9. doi: 10.1161/01.CIR.0000070954.00271.13. Epub 2003 May 19. PMID 12756158
- [Background] Sun T, Hu J, Yin Z, Xu Z, Zhang L, Fan L, Zhuo Y, Wang C. Low serum paraoxonase1 activity levels predict coronary artery disease severity. Oncotarget. 2017 Mar 21;8(12):19443-19454. doi: 10.18632/oncotarget.14305. PMID 28038449
- [Background] Shen Y, Ding FH, Sun JT, Pu LJ, Zhang RY, Zhang Q, Chen QJ, Shen WF, Lu L. Association of elevated apoA-I glycation and reduced HDL-associated paraoxonase1, 3 activity, and their interaction with angiographic severity of coronary artery disease in patients with type 2 diabetes mellitus. Cardiovasc Diabetol. 2015 May 13;14:52. doi: 10.1186/s12933-015-0221-4. PMID 25964115
- [Background] Gur M, Aslan M, Yildiz A, Demirbag R, Yilmaz R, Selek S, Erel O, Ozdogru I. Paraoxonase and arylesterase activities in coronary artery disease. Eur J Clin Invest. 2006 Nov;36(11):779-87. doi: 10.1111/j.1365-2362.2006.01727.x. PMID 17032345
- [Background] Ragab M, Hassan H, Zaytoun T, Refai W, Rocks B, Elsammak M. Evaluation of serum neopterin, high-sensitivity C-reactive protein and thiobarbituric acid reactive substances in Egyptian patients with acute coronary syndromes. Exp Clin Cardiol. 2005 Winter;10(4):250-5. PMID 19641675
- [Background] Walter MF, Jacob RF, Jeffers B, Ghadanfar MM, Preston GM, Buch J, Mason RP; PREVENT study. Serum levels of thiobarbituric acid reactive substances predict cardiovascular events in patients with stable coronary artery disease: a longitudinal analysis of the PREVENT study. J Am Coll Cardiol. 2004 Nov 16;44(10):1996-2002. doi: 10.1016/j.jacc.2004.08.029. PMID 15542282
- [Background] Azarsiz E, Kayikcioglu M, Payzin S, Yildirim Sozmen E. PON1 activities and oxidative markers of LDL in patients with angiographically proven coronary artery disease. Int J Cardiol. 2003 Sep;91(1):43-51. doi: 10.1016/s0167-5273(02)00595-8. PMID 12957728
- [Background] Altiparmak IH, Erkus ME, Sezen H, Demirbag R, Gunebakmaz O, Kaya Z, Sezen Y, Asoglu R, Dedeoglu IH, Neselioglu S, Erel O. The relation of serum thiol levels and thiol/disulphide homeostasis with the severity of coronary artery disease. Kardiol Pol. 2016;74(11):1346-1353. doi: 10.5603/KP.a2016.0085. Epub 2016 May 25. PMID 27221962
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Background] Antman EM, Cohen M, Bernink PJ, McCabe CH, Horacek T, Papuchis G, Mautner B, Corbalan R, Radley D, Braunwald E. The TIMI risk score for unstable angina/non-ST elevation MI: A method for prognostication and therapeutic decision making. JAMA. 2000 Aug 16;284(7):835-42. doi: 10.1001/jama.284.7.835. PMID 10938172
- [Background] Fox KA, Dabbous OH, Goldberg RJ, Pieper KS, Eagle KA, Van de Werf F, Avezum A, Goodman SG, Flather MD, Anderson FA Jr, Granger CB. Prediction of risk of death and myocardial infarction in the six months after presentation with acute coronary syndrome: prospective multinational observational study (GRACE). BMJ. 2006 Nov 25;333(7578):1091. doi: 10.1136/bmj.38985.646481.55. Epub 2006 Oct 10. PMID 17032691